CLINICAL TRIAL: NCT03359629
Title: Accuracy Evaluation of Glucometry Monitor Developed by Spectrophon LTD
Brief Title: Spectrophon LTD Glucometry Monitor Accuracy
Status: Completed | Type: Observational
Sponsor: Tirat Carmel Mental Health Center (Other Government)
Collaborators: Ariel University (Other)
Responsible Party: Principal Investigator, Anatoly Kreinin, MD, PHD, Clinical Assistant Professor, Tirat Carmel Mental Health Center
Other Study IDs: SGM-1
Record Dates: First submitted 2017-11-23; First posted 2017-12-02 (Actual); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2018-11

CONDITIONS: Glucose Metabolism Disorders; Diabetes Mellitus
Keywords: Spectrophon; Glucose; Biosensor; Non-invasive testing
MeSH Terms: conditions — Glucose Metabolism Disorders; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Spectrophon Glucometry Monitor — Wearable smartwatch with integrated non-invasive glucose detection system
Device: YSI 2300 Stat Plus — Reference commercial glucometer

SUMMARY:
Diabetes mellitus (or diabetes) is a chronic, metabolic disease characterized by elevated levels of blood glucose. Patients with diabetes need to monitor their blood glucose level several times a day to control their medical state. Modern biosensors have become a promising solution for non-invasive blood glucose measurements. This study aims to validate the efficacy and the accuracy of Glucometry Monitor (NIGM) developed by Spectrophon LTD incorporated in smart watches.

Method Participants will use Spectrophon biosensors to non-invasively estimate the level of glucose in blood. Blood will also be collected and the glucose level will be checked with commercially available blood glucose analyzers . All sets of data will be compared to estimate the accuracy of measurements of Spectrophon NIGM

DETAILED DESCRIPTION:
Diabetes is a chronic, life-long disease that represents a major public health challenge at a world level (Matthews et al 1985). It is important to note that diabetes is common among mentally ill patients, especially among patients with schizophrenia that are treated with new generation antipsychotic drugs (Nielsen et al 2010, Vancampfort et al 2016).

To maintain blood glucose level homeostasis, repeated blood glucose testing is needed. The vast majorities of currently available methods for blood glucose testing are invasive and cause discomfort for patients. However, biosensors have recently become a promising solution for non-invasive glucose blood testing (Bandodkar et al 2014; Zhang et al 2015). Spectrophon LTD has developed a technology that allows measurement of even the smallest amounts of various compounds contained in sweat. Using unique algorithm developed by Spectrophon LTD, these data provides the possibility of evaluating the levels of chemicals in the bloodstream. Based on this technology, Spectrophone LTD has developed a glucometer biosensor that is able to non-invasively detect the blood glucose level. This glucometer biosensor can be easily incorporated into most commercially available smartwatches. Development of this technology will allow real-time, non-invasive measurement of blood glucose level and will dramatically facilitate effective treatment of diabetes. In addition, this technology will enable monitoring of glucose levels in patients with mental disorders that will facilitate the early detection of metabolic syndrome.

Study Design: this naturalistic study will examine the accuracy of Spectrophon NIGM incorporated in smart watch Samsung Gear S2 that non-invasively and indirectly detect the level of glucose in human blood. The study will be held in Maale Carmel Mental Health Center (MCMHC). Adult participants (n=200) will be recruited for the study from the staff of MCMHC (including doctors, nurses and administrative workers; no psychiatric in-patients will be recruited for the study). In parallel to glucose measurements with NIGM, blood will be collected and the glucose level will be checked using commercially available blood glucose analyzers.

The participants will be able to select between two options for blood collection:

The first option: intravenous cannula (Venflon) will be inserted in cubital vein and blood will be collected twice in the beginning and at the end of the procedure (within 1-3 hours) and checked for the glucose level with commercially available blood glucose analyzers.

The second option: The blood will be collected twice from the cubital vein at the beginning and at the end of the procedure (within 1-3 hours) and checked for the glucose level using commercially available blood glucose analyzers .

The measurements will be performed twice: before meal (subject should be in fasting state) and after meal with one hour interval between two measurements.

The results of the measurements of the NIGM will be compared to the results obtained from commercially available blood glucose analyzers.

The application automatically saves every measurement into archive. To better control the process, the manual fixation of data obtained by NIGM is performed.

ELIGIBILITY:
Inclusion Criteria:

* must be between ages 18 and 75
* must be able to sign informed consent form.

Exclusion Criteria:

* Acute psychotic state
* Hepatitis
* HIV
* Tuberculosis
* Haemophilia and other serious coagulation disorders
* Significant impaired venous access
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Israeli and non-israeli citizens of age 18-75.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly Kreinin, MD, PHD, Principal Investigator — Bruce Rappaport Medical Faculty, Technion, Haifa, Israel
Locations (1):
- Tirat Carmel Mental Health Center, Tirat Carmel, Haifa District, Israel

RESULTS

PARTICIPANT FLOW:
Groups:
- Blood Collection (Healthy Individuals): Participants's blood was collected and measured for glucose level before and after food intake
- Blood Collection (Diabetic Patients): Participants's blood was collected and measured for glucose level
Period: Overall Study
Arm/Group | Blood Collection (Healthy Individuals) | Blood Collection (Diabetic Patients)
Started | 200 | 10
Completed | 200 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blood Collection (Healthy Individuals) | Blood Collection (Diabetic Patients) | Total
Number analyzed (Participants) | 200 | 10 | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 188 | 7 | 195
  >=65 years | 12 | 3 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 7 | 121
  Male | 86 | 3 | 89
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 200 | 10 | 210

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Measurements With < 15% Error
Description: Difference in measurements of blood glucose level obtained using Spectrophon glucometry monitor and commercially available glucose analyser YSI 2300
Time Frame: 1-3 hours
Measure: Number; unit: Percentage of measures with error <15%
Arm/Group | Blood Collection (Healthy Individuals) | Blood Collection (Diabetic Patients)
Number analyzed (Participants) | 200 | 10
Percentage of measures with error <15%
  Algorithm 1.7 | 95.25 | 100
  Algorithm 1.6 | 94.5 | 100

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Blood Collection (Healthy Individuals) | Blood Collection (Diabetic Patients)
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/10
Other Adverse Events (participants affected / at risk) | 0/200 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT03359629/Prot_SAP_000.pdf